CLINICAL TRIAL: NCT05402579
Title: Diabetic Ketoacidosis From New SGLT2i: Can Genomics Estimate Risk (DaNGER)
Brief Title: Diabetic Ketoacidosis From New SGLT2i: Can Genomics Estimate Risk
Acronym: DaNGER
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Unity Health Toronto (Other); University Health Network, Toronto (Other); Sault Area Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 3737
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Type 2; DKA; Diabetic Ketoacidosis
Keywords: DKA; SGLT2i; Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: None Retained — Genetic samples will be collected using a DNA saliva collection kit (Oragene: OG-510) and will be sent for genome-wide genotyping to The Centre for Applied Genomics in The Hospital for Sick Children (SickKids)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with type 2 diabetes mellitus who were hospitalized with SGLT2 inhibitor-associated DKA (60 cases).
  Interventions: Genetic: Genomic analysis
- Controls: There are two sources for controls. [1] Patients hospitalized at one of the participating hospitals who were on an SGLT2i and do not have DKA. [2] Population controls using publicly available data from the Canadian Longitudinal Study on Aging (CLSA) database (1000 controls via CLSA).
  Interventions: Genetic: Genomic analysis

INTERVENTIONS:
Genetic: Genomic analysis — Genetic samples will be collected using a DNA saliva collection kit (Oragene: OG-510) and will be sent for genome-wide genotyping to The Centre for Applied Genomics in The Hospital for Sick Children (SickKids)

SUMMARY:
Sodium glucose co-transporter 2 (SGLT2) inhibitors have revolutionized care for people living with type 2 diabetes mellitus (T2DM). They reduce a person's risk of heart failure, renal failure, myocardial infarction, stroke, cardiovascular mortality, and potentially all-cause mortality. Remarkably, some of these benefits also extend to people who do not have T2DM. While the benefits of SGLT2 inhibitors are impressive, there is one life-threatening side effect associated with their use: diabetic ketoacidosis (DKA). The ability to predict which patients are at highest risk of DKA is needed to sufficiently mitigate this risk. Moreover, considering the impressive benefits of SGLT2 inhibitors, identifying patients at the lowest risk of SGLT2 inhibitor-associated DKA is also important so that providers do not overestimate risk in those who stand to benefit most.

Advances in genomic technologies and related analyses have provided unprecedented opportunities to bring genomics-driven precision medicine initiatives to the forefront of clinical research. Leading these developments has been the progress made by genome-wide association studies (GWAS) due to decreasing genotyping costs, and consequently, the ability to routinely study large numbers of patients. These approaches allow for systematic screening of the genome in an unbiased manner and have accelerated the discovery of genetic variants and novel biological processes that contribute to the development of adverse treatment outcomes.

By using innovative approaches, which harness large cohorts of population controls, sample size limitations that are associated with rare adverse drug reactions such as SGLT2 inhibitor-associated DKA can be overcome. The DANGER study represents a highly innovative new direction wherein partnership among basic science researchers and computational biologists will lead to the application of genomic techniques to identify genetic variants that may be associated with SGLT2 inhibitor-associated DKA.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for participation in this study, a participant must meet each of the following criteria:

1. Be 18 years or older and have a diagnosis of type 2 diabetes mellitus.
2. Have been admitted to hospital with SGLT2 inhibitor-associated DKA (cases) or admitted to hospital on an SGLT2 inhibitor and not have DKA (controls).
3. Be able to provide written consent (or, if patient is unable, have a substitute decision maker [SDM] available).

Exclusion Criteria:

A participant will be ineligible for participation in this study if he or she satisfies any one or more of the following criteria:

1. Diagnosis of type 1 diabetes mellitus.
2. Unable to spit 10mL into a vial.
3. A first degree relative has already been recruited into the study.
4. Had an alcohol binge before admission
5. Had prolonged fasting (>48 hours) prior to hospital admission
6. Recently stopped their insulin (within the past 7 days prior to hospital admission)

Our study will not include children or pregnant women because SGLT2 inhibitors are not approved for use in either patient population.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases: Patients with type 2 diabetes mellitus who were hospitalized with SGLT2 inhibitor-associated DKA will be eligible for inclusion in our study.
  Controls: There are two sources for controls. [1] Patients hospitalized at one of the participating hospitals who were on an SGLT2i and do not have DKA. [2] Population controls using publicly available data from the Canadian Longitudinal Study on Aging (CLSA) database.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Identification of genomic variants associated with an increased risk of SGLT2 inhibitor-associated DKA | One year
  Genetic ancestry will be calculated using principal component analyses and outliers will be removed. GWAS will be performed with SAIGE, including genetic ancestry and the relevant clinical/demographic variables as covariates, to identify genetic variants associated with SGLT2 inhibitor-associated DKA.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Health Centre (Unity Health Toronto), Toronto, Ontario
  - Toronto General Hospital (University Health Network), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No